CLINICAL TRIAL: NCT04851925
Title: MR-Fingerprinting for the Prediction of the Response of Vestibular Schwannomas to Gamma Knife Radiosurgery
Brief Title: MR Fingerprinting for Vestibular Schwannomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Josa M Frischer, MD, PhD, Principal Investigator, Medical University of Vienna
Other Study IDs: EK2451/2020
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Vestibular Schwannoma
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MR Fingerprinting — Specific Magnetic Resonance Imaging protocol

SUMMARY:
MR Fingerprinting (MRF) will be performed in patients who will be treated with Gamma Knife radio surgery for a vestibular schwannoma before the intervention. Fifty patients will be included with a vestibular schwannoma of minimum 1cm in size. During follow-up, response of the tumor to radiosurgery will be evaluated for each patient with MRI. The aim of the study is to find patterns of vestibular schwannomas in MRF data which correlate with the type of response to radio surgery, i.e. tumor control after radiosurgery, further tumor growth despite radiosurgery, cystic transformation after radiosurgery.

ELIGIBILITY:
Inclusion Criteria: Planned Gamma Knife radiosurgery for vestibular schwannoma of minimum 1cm in size -

Exclusion Criteria: Vestibular Schwannoma of less than 1cm in size. Other a priori treatment than Gamma Knife radiosurgery

-

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with vestibular schwannoma of minimum 1cm, who will undergo Gamma Knife radiosurgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Tumor control | 3 years
  Number of patients without further growth of the tumor on follow-up MRI after radiosurgery
Tumor growth | 3 years
  Number of patients with growth of the tumor on follow-up MRI after radiosurgery
Cystic transformation | 3 years
  Number of patients with cystic transformation of the tumor on follow-up MRI after radiosurgery

CONTACTS AND LOCATIONS:
Overall Officials: Josa Frischer, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No